CLINICAL TRIAL: NCT06681623
Title: A Single-Center, Prospective Cohort Study to Characterize the Safety and Efficacy of Ublituximab in Older Adults With Relapsing Forms of Multiple Sclerosis (RMS)
Brief Title: A Single-Center Study to Characterize the Safety and Efficacy of Ublituximab in Older Adults With Relapsing Forms of Multiple Sclerosis (RMS)
Status: Recruiting | Type: Observational
Sponsor: Neurology Center of New England P.C. (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00078205
Record Dates: First submitted 2024-10-28; First posted 2024-11-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis, Relapsing Forms of Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ublituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Ublituximab — Drug: ublituximab

SUMMARY:
The purpose of this study is to evaluate the safety of ublituximab use in the older MS adult population, as measured by incidence of infection rate

DETAILED DESCRIPTION:
This study is being done to see how safe and effective ublituximab is when given to older adult patients for their RMS. Since RMS patients over age 55 were excluded from previous clinical studies that studied the safety and efficacy of ublituximab, this study is designed to better understand how well this drug is tolerated in RMS patients between the ages of 55-80 years.

Primary endpoints include:

* Incidence of infection rate from Baseline to Month 24/EOS (including UTI and other active acute, opportunistic and/or chronic infection)
* Incidence of TEAS/SAEs from Baseline to Month 24 with consideration to nature, severity, and occurrence rate of AEs

Approximately 20 participants are expected to be enrolled. Participation in this study will last approximately 24 months and will include approximately 6 study visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Aged 55-80 years old
* Diagnosis of RMS according to the 2017 Revised McDonald criteria
* Anticipated to begin treatment with or newly treated with ublituximab (within 6 months prior to study entry) according to the local label

Exclusion Criteria:

* Active participation in an interventional clinical trial for MS
* Received initial dose of ublituximab more than 6 months prior to study entry
* History of life-threatening infusion reaction on any anti-CD20 therapy
* Evidence of clinically significant chronic or ongoing active viral, bacterial, or fungal infectious disease requiring long term systemic treatment, or any history of recurrent infection within 6-12 months prior to initiation of ublituximab

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects meeting protocol-specified criteria will be recruited from the Neurology Center of New England P.C.'s internal patient database
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection (including UTI and other active acute, opportunistic and/or chronic infection) | From Baseline to Month 24/End of Study
  Incidence of infection rate from Baseline to Month 24/End of Study
Incidence of treatment-emergent adverse events (TEAEs)/serious adverse events (SAEs) | From Baseline to Month 24/End of Study
  Incidence of TEAEs/SAEs from Baseline to Month 24/End of Study

SECONDARY OUTCOMES:
Total number of new and/or enlarging T2 lesions on all available brain MRI scans | From Baseline to Month 24/End of Study
  Change from Baseline to Month 24/End of Study in total number of new and/or enlarging T2 lesions on all available brain MRI scans
Functional Assessment (Expanded Disability Status Scale (EDSS)) | From Baseline to Month 24/End of Study
  Change from Baseline to Month 24/End of Study in EDSS
Multiple Sclerosis Impact Scale (MSIS-29) | From Baseline to Month 24/End of Study
  Change from Baseline to Month 24/End of Study in Multiple Sclerosis Impact Scale (MSIS-29)
Absolute lymphocyte count (ALC) | From Baseline to Month 24/End of Study
  Change from Baseline to Month 24/End of Study in ALC
Immunoglobulin levels | From Baseline to Month 24/End of Study
  Change from Baseline to Month 24/End of Study in immunoglobulin levels
Functional Assessment (Timed 25-Foot Walk Test (T25-FW)) | From Baseline to Month 24/End of Study
  Change from Baseline to Month 24/End of Study in T25-FW

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Center of New England P.C., Foxborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided